CLINICAL TRIAL: NCT03362554
Title: Identification of New Biomarkers of Insulin Resistance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Teagasc (Industry)
Responsible Party: Principal Investigator, Francoise Koumanov, Lecturer, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC-FH1158
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Insulin Resistance; Diabetes Mellitus, Type 2; Inflammation; Gastrointestinal Microbiome
Keywords: Insulin; Glucose; Rab3
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Controlled diet and exercise.
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Controlled diet and exercise. — The intervention will involve 3 weeks of a diet and exercise program designed to cause a net energy decrease of 7000 kcal/week compared to habitual behaviour. This will be achieved through:
  * Five exercise sessions per week at 70% VO2 max, using 400 kcal per session.
  * Reduction of their standard diet by 5000 kcal per week
  Before and after this intervention period participants will take part in a trial day which includes measurement of body composition (using DEXA) and blood sugar control (oral glucose tolerance test). Samples of blood, adipose, skeletal muscle and faeces will also be taken.
  Arms: Intervention

SUMMARY:
Diabetes is a chronic metabolic disease affecting 415 million people worldwide, 90% of cases are type 2 which is frequently associated with obesity and a sedentary lifestyle. In healthy individuals, insulin stimulates increased cell surface expression of a glucose transporter (GLUT4) in muscle and fat tissue. This prevents blood sugar levels becoming dangerously high by taking sugar into the muscle and fat cells. Loss of this response ('insulin resistance') frequently occurs before the development of type 2 diabetes. Understanding the cell biology of insulin resistance is necessary to develop more effective treatments for this condition and prevent further cases of type 2 diabetes. Previous work showed that this movement of GLUT4 is dependent on a small protein called Rab3 which is downregulated in insulin resistance. Rab3 protein levels are also sensitive to inflammation, a state that is exacerbated by obesity.

In order to examine whether Rab3 is an early biomarker of insulin resistance, we aim to measure the levels of this protein and its interactors in fat and muscle samples from insulin resistant individuals. It has been shown that insulin sensitivity can be improved with an intervention as short as three weeks when net energy intake is sufficiently reduced. Therefore, by taking the same measurements before and after this three week intervention we can observe any improvements in Rab3 expression and insulin sensitivity at a cellular level.

There is also evidence for an effect of the gut microbiome on insulin sensitivity so we will measure any changes that take place in the gut microbiome following this intervention, which can be determined from faecal samples taken before and after the three weeks.

DETAILED DESCRIPTION:
Diabetes is a chronic metabolic disease affecting 415 million people worldwide and 3.5 million people in the UK, with ninety percent suffering from type 2 diabetes. Type 2 diabetes is characterised by the inability of muscle and fat tissues to adequately respond to physiological levels of insulin (peripheral tissue insulin resistance), and to restore the normal levels of sugars in the bloodstream. Insulin resistance may occur prior to the development of type 2 diabetes and has been shown to be strongly linked to lifestyle and to obesity, although the underlying mechanisms are incompletely resolved. A defining characteristic of insulin resistance is abnormal glucose transport as a result of decreased cell surface expression of the glucose receptor GLUT4. In healthy adipose and skeletal muscle this receptor is trafficked to the cell surface in response to an insulin stimulus. We have shown that this translocation to the cell membrane requires the protein Rab3, and expression levels of this protein are reduced in cell models of insulin resistance.

We hypothesise that this downregulation of Rab3 is associated with the development of insulin resistance and its activity would increase following the restoration of insulin sensitivity. The primary aim of this study is to examine the effect on Rab3 levels and GLUT4 trafficking of a diet and exercise intervention that has been previously shown to increase insulin sensitivity. Additionally, the gut microbiome will be studied before and after the intervention to determine any relationship to insulin sensitivity. Recent evidence suggests the microbiome has a significant role in the development of insulin resistance through a number of potential mechanisms. Infusion of microbiota from lean donors has been shown to result in improved insulin sensitivity in male recipients with metabolic syndrome, with concomitant increases in the prevalence of butyrate-producing intestinal microbiota. Exercise is associated with greater microbial diversity, including increases in butyrate-producing microbes. No study to date has monitored insulin sensitivity and microbiota composition before and after an exercise and diet intervention, and so this will lead to a better understanding of the mechanisms that lead to insulin resistance and subsequently type 2 diabetes.

The study participants will include males and females aged between 40-65 years who fit the criteria for inclusion. After monitoring of normal daily activities for 7 days, volunteers will reduce their calorie intake by 5000 kcal/week and take part in 5 weekly exercise sessions for 3 weeks. Participants will attend one session of laboratory testing before and one after this period which will take place at the University of Bath. This intervention should be sufficient to improve insulin sensitivity and allow us to study the cellular changes that will have taken place during this time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 40-65
* BMI ≥25 to ≤ 40 kg/m2
* Physical activity level <1.75 (daily average)
* Waist size >80 cm (female) or >94 cm (male)
* Weight stable for >3 months

Exclusion Criteria:

* Inability to undertake exercise as determined by PAR-Q
* Diagnosed diabetes
* Ongoing or planned lifestyle changes (diet/exercise)
* Recent large shift in bodyweight (>2.5%) within the last 3 months?
* Smoker (or having ceased <6mo ago)
* Metabolic disorders
* Hypertension defined as >160/100
* Use of anti-inflammatory medication: NSAIDs
* Cardiovascular disease
* Any bleeding disorder or taking anticoagulant medication
* Use of antibiotics within the last three months
* Use of pro/pre-biotics within one month of first trial day.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity | 120 min (change after 3 weeks)
  Response to oral glucose tolerance test

SECONDARY OUTCOMES:
Rab3 protein expression | Change after 3 weeks
  Levels of Rab3 in adipose and muscle samples
GLUT4 pathway protein expression | Change after 3 weeks
  Expression levels of GLUT4 pathway proteins in adipose and muscle samples
Metabolic markers | Change after 3 weeks
  Levels of circulating metabolic markers implicated in insulin resistance
Inflammatory markers | Change after 3 weeks
  Levels of circulating inflammatory cytokines
Gut microbiome | Change after 3 weeks
  Species of microorganisms present in fecal samples
Body composition | Change after 3 weeks
  Assessed by whole body DEXA scan
Waist circumference | Change after 3 weeks
Body mass | Change after 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Koumanov, PhD, Principal Investigator — University of Bath
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiabetesUK, Facts and Stats. 2016: https://diabetes-resources-production.s3-eu-west-1.amazonaws.com/diabetes-storage/migration/pdf/DiabetesUK_Facts_Stats_Oct16.pdf.
- [Background] Kahn BB, Flier JS. Obesity and insulin resistance. J Clin Invest. 2000 Aug;106(4):473-81. doi: 10.1172/JCI10842. No abstract available. PMID 10953022
- [Background] Koumanov F, Pereira VJ, Richardson JD, Sargent SL, Fazakerley DJ, Holman GD. Insulin regulates Rab3-Noc2 complex dissociation to promote GLUT4 translocation in rat adipocytes. Diabetologia. 2015 Aug;58(8):1877-86. doi: 10.1007/s00125-015-3627-3. Epub 2015 May 30. PMID 26024738
- [Background] Walhin JP, Dixon NC, Betts JA, Thompson D. The impact of exercise intensity on whole body and adipose tissue metabolism during energy restriction in sedentary overweight men and postmenopausal women. Physiol Rep. 2016 Dec;4(24):e13026. doi: 10.14814/phy2.13026. PMID 28039399
- [Background] Utzschneider KM, Kratz M, Damman CJ, Hullar M. Mechanisms Linking the Gut Microbiome and Glucose Metabolism. J Clin Endocrinol Metab. 2016 Apr;101(4):1445-54. doi: 10.1210/jc.2015-4251. Epub 2016 Mar 3. PMID 26938201
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Campbell SC, Wisniewski PJ 2nd. Exercise is a Novel Promoter of Intestinal Health and Microbial Diversity. Exerc Sport Sci Rev. 2017 Jan;45(1):41-47. doi: 10.1249/JES.0000000000000096. PMID 27782912